CLINICAL TRIAL: NCT02622360
Title: Speech and Short-term Memory Functions in Dyslexia: a Combined MEG and EEG Study
Acronym: SMeDy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Teija Kujala, Prof., University of Helsinki
Other Study IDs: 12345
Record Dates: First submitted 2015-11-11; First posted 2015-12-04 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — extraction of DNA from whole blood samples or saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dyslexia: Individuals with confirmed dyslexia.
- Control: Healthy control subjects.

SUMMARY:
Developmental dyslexia is a highly heritable disorder in which reading skills are compromised despite normal intelligence and appropriate reading instruction. Reading problems in dyslexia are thought to primarily originate from weak speech sound representations or poor phonological skills. Dyslexia has also been associated with short-term or working memory dysfunctions. The current study will address the presence of these problems in dyslexic adults by the means of recording auditory and audio-visual mismatch negativity (MMN) and its magnetic counterpart (MMNm) to determine neural speech sound discrimination, representations and integration of seen and heard language. In addition to analyzing neural processing of syllables or (pseudo-)words, a new approach to MEG acquisition and analysis to characterize the neural responses during comprehension of complex real-life speech will be used. Furthermore, reading, phonological and cognitive skills of these participants will be determined with a neuropsychological test battery. The associations between the neural, neuropsychological and genetic measures will be studied. This project will illuminate the nature of neurocognitive dysfunctions in dyslexia and their relationship with genes.

DETAILED DESCRIPTION:
1. Background

   Developmental dyslexia is the most prevalent learning disorder impairing reading skill even in individuals having normal intelligence and full availability of education (Lyon et al., 2003). It is highly heritable, and several candidate genes contributing to dyslexia have been identified (Scerri & Schulte-Körne, 2010). A wide range of deficits have been associated with dyslexia, but according to the most prevalent theory its major cause is impaired phonological processing (Ramus, 2001). The MMN, the generators of which overlap with brain areas reported to have anatomical abnormalities in dyslexia, has supported this notion. Diminished MMN amplitudes have systematically been reported in dyslexics for certain speech and non-speech sound features (for a review Kujala & Näätänen, 2001). These effects were even found in children and infants having an inherited risk for dyslexia (Leppänen et al., 2002; Lovio et al., 2010). Furthermore, a recent study in our group has shown that dyslexic children have problems in forming memory traces for words (Kimppa et al., in prep.), whereas both the auditory system of normal-reading adults (Shtyrov et al., 2010) and children (Kimppa et al., in prep.) was shown to rapidly form representations for novel words.

   It was recently suggested that phonological deficits in dyslexia can occur due to impairments in different steps of sound processing. According to this theory, dyslexic individuals can be divided into different subgroups. Ramus and colleagues (2013) suggested that dyslexic individuals show an impairment in phonological representations or at later processing stages as an impairment in phonological skills.

   The current project will utilize combined electroencephalographic (EEG) and magnetoencephalographic (MEG) recordings and neuropsychological and perceptual testing in order to determine how impaired phonological neural representations vs. phonological skills contribute to dyslexia. Defined as time-locked changes to external stimuli in EEG and magnetoencephalogram MEG, event-related potentials (ERPs) and event-related fields (ERFs), respectively, could provide an objective index of information processing in the human brain. Both EEG and MEG methods offer a high temporal resolution. The benefit of MEG is offered by a more exact localization of the activated neural sources due to a diminished effect of distortions caused by the skull and tissue than in the process of EEG source localization. It will complement and add more specific information to dyslexia ERP research additional to the previous studies that were mostly conducted with EEG. For a summary of dyslexia studies conducted with MEG, see the review from Salmelin (2007).

   Neural responses recorded with EEG and MEG have widely been used both in the service of basic research and clinically-oriented research. During the recent years, a cortical response called the mismatch negativity (MMN) has been in intensive use in investigating auditory perception and its deficits. MMN is an ERP component elicited by any change in some repetitive aspect of auditory stimulation, peaking at 100-200 ms from change onset and detectable both electrically (MMN) and magnetically (MMNm). It was suggested that MMN provides an index of the auditory sensory ("echoic") memory and automatic (involuntary) change-detection. It also reflects native-language specific speech-sound memory traces (Näätänen et al., 1997). MMN is elicited even when the subject is not attending the auditory stimuli. Therefore, it has been popular in investigating a variety of patient groups during the recent years (for reviews, see Näätänen et al., 2007; Kujala et al., 2007).

   In addition to the processing of syllables or (pseudo-)words, the neural activity during comprehension of complex real-life speech by recording single-trial MEG will be characterized. A model-free analysis method investigates inter-subject correlations (ISC) between individuals with and without dyslexia. This approach will give insight about auditory processing characteristics in a more natural condition. The method of ISC has been proven viable in research during natural conditions, e.g. movie watching or listening to music, mainly using functional magnetic resonance imaging (fMRI). It has been introduced by Hasson and colleagues in 2004, who found that brain regions synchronize between subjects during movie viewing. In MEG, this approach has only been used scarcely (e.g. Lankinen et al., 2014; Suppanen, 2014; Thiede, 2014). However, it confirms and complements the results from fMRI research. In language research, temporal correlations that were investigated with the ISC method, have only been reported in resting state networks in children with reading difficulties (Dimitriadis et al., 2013). The results confirm findings from fMRI studies. Thus, the method offers new, promising insights into the neural underpinnings of dyslexia.

   Developmental dyslexia is a heritable disorder with polygenic origin. Several candidate genes have been detected in the recent years (Kere, 2014 for a review), associated with functions of neuronal migration and auditory processing. However, the connection between the auditory responses of the brain and the genetic cause of the disorder has not been confirmed yet. More research on the connections between the genetic and neural markers of dyslexia is needed in order to verify different existing hypotheses.

   Previous activity

   Research in the experimenters group has shown that at group level, cortical low-level discrimination of sounds and speech sounds is impaired in dyslexia (Kujala, 2007 for a review). This was reflected in diminished MMN responses (e.g., Kujala et al., 2006; Schulte-Körne et al., 1998; Neuhoff et al., 2012) and in enhancements of MMNs as a result of dyslexia intervention (Kujala et al., 2001; Lovio et al., 2012). These results suggest a strong connection between this neural response and dyslexia. Furthermore, the investigators' results suggest weak associations between the neural representations of speech sounds and written letters in the brains of dyslexics (Mittag et al., 2013), which could reflect deficits in phonological skills in dyslexia. Furthermore, studies carried out in the current research group have lead to the identification of candidate genes of dyslexia (e.g. Hannula-Jouppi et al., 2005; Schumacher et al., 2006). In a recent review, nine genes and four gene loci have been listed in a summary of genetic loci associated with developmental dyslexia (Kere, 2014). Some candidate genes were shown to be linked with axonal connections and others with neuronal migration functions.
2. Objectives and methods

This study aims at determining neurocognitive underpinnings of dyslexia and their connection with genes. The target neural processes impaired in different subgroups of dyslexic individuals involve phonological representations vs. phonological skills. Phonological representations are reflected in the low-level discrimination of speech sounds, whereas phonological skills can be mirrored in audiovisual integration of written and spoken letters. With neuropsychological tests, it will be determined which participants have primarily weak speech representations or poor phonological skills. It is hypothesized that participants with weak phonological representations have diminished MMN/MMNm responses. However, participants who do not have these problems, but instead have poor phonological skills, are expected to have normal-like MMN/MMNm responses but deficient responses reflecting audiovisual integration, such as no difference in effects of printed text versus nonsense visual material on early auditory speech discrimination. These two types of dyslexic groups are hypothesized to have alterations in partly different dyslexia candidate genes.

Auditory processing in the brain under more complex, real-world conditions will be investigated using single-trial MEG during presentation of natural speech sounds. It is expected that the synchronized brain activity differs between the dyslexic and control group. Specifically, it is expected that dyslexic subjects show decreased synchrony in the left temporoparietal cortex (Temple, 2002). Single-trial data could furthermore show a connection to genes, as suggested by Giraud and Ramus (2013), who hypothesized that a disruption of auditory cortical oscillations modifies the access to phonological representations.

Dyslexia is known to be associated with several candidate genes (for a review, see Kere, 2014). The candidate genes are associated with language skills and with the brain's ERPs. The gene research in cooperation with Prof. Juha Kere's laboratory in Folkhälsan research centre in Biomedicum, Helsinki or Karolinska Institutet, Stockholm, will aim at proofing the connection between dyslexia candidate genes and neural event-related activity of the brain to pseudoword stimuli.

Stimuli and procedure

MMN and MMNm responses to sound changes in pseudoword /tata/ (vowel, vowel duration, and syllable frequency changes) will be recorded while participants attend a movie or see concurrent visually-presented pseudoword stimuli. During the auditory condition, subjects will watch a silenced movie while being presented frequent "standard" stimuli, namely a pseudoword (/tata/) and infrequent "deviant" (see below) auditory stimuli. The task is to attend the movie and to ignore the background sounds. The audiovisual condition includes the same pseudoword stimuli, but instead of watching a movie, subjects will see the written letters of the presented pseudoword or a scrambled picture of the pseudoword letters. Distractors, such as counting deviant stimuli or different shapes and colours of the visual stimulus, will be given as the main task to the participants. They will be instructed to ignore the sounds.

The pseudoword stimuli are as follows:

* standard: /tata/
* vowel deviant: /tato/
* frequency deviant - higher frequency in the 2nd syllable
* duration deviant: /tataa/ - 2nd syllable twice as long as in the standard

The stimuli will be presented in a combined multi-feature and oddball design (Näätänen et al., 2004). All deviant types will be presented in the same sequence with 1-4 standards between each successive 2 deviants.

In addition to recording MMNm responses, a single-trial, continuous recording of brain activity for a real-world stimulus will be recorded. Approximately 8 min of natural speech (Finnish speaker) will be presented to both groups with the task of mere listening and keeping the eyes open. A recording of 8 min during rest with eyes open will complete the addition.

In order to examine differences in general cognitive abilities and performance profile between groups, the participants will undergo behavioural tests. Dyslexia characteristics will be assessed with parts of the Nevala dyslexia test (Nevala et al., 2006). General and performance Intelligence Quotient (IQ) as well as phonological and working memory will be tested using the Wechsler Intelligence Scale (WAIS-III; Wechsler, 1997a) and subtests of Wechsler Memory Scale (WMS-III; Wechsler, 1997b). Phonological naming will be assessed with the rapid alternate stimulus naming (RAS) test for speed and accuracy (Wolf, 1986). These or corresponding neuropsychological tests will be executed in max. 2 hours in an independent test session from the MEG session.

Additionally, saliva or blood samples (2x9 ml blood) will be collected by a trained nurse after subject's approval. DNA will be extracted from these samples and stored in Folkhälsan research centre in Juha Kere's laboratory. The DNA analysis focuses on any related candidate genes in their different variants using DNA sequencing techniques to determine the genotypes (Taqman, Sequenom). Possible links between the electric and magnetic activity of the brain and candidate genes for dyslexia are searched for.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 year old
* Finnish-speaking
* right-handed
* normal hearing and normal or corrected-to-normal vision
* dyslexic (if not, it is possible to participate as a control participant)

Exclusion Criteria:

* known neurological or psychiatric diseases
* history of alcohol or drug abuse
* metal in the body

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 Finnish healthy adult subjects aged 18-45 will be tested, around half of who have a developmental dyslexia. Prior to the study, subjects are given "Written investigation information" after which the subjects may participate in the study by signing the "Written informed consent".
  Participants in the dyslexia group are required to have a prior diagnosis of dyslexia as an inclusion criterion. Groups will be matched for gender, age and educational level. The participation to the experiment is on voluntary basis after announcement through different channels, e.g. via email lists. All experiments will be carried out according to the Declaration of Helsinki.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2017-04 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Magnetic mismatch negativity brain responses to speech sound changes | 2 hours

SECONDARY OUTCOMES:
Magnetoencephalographic amplitude envelope inter-subject correlation during listening to complex real-life speech | 2 hours
Event-related brain responses to pseudowords | first 25% and last 25% of the measurement time (total 2 hours)
Correlation of event-related brain responses to susceptibility genes for dyslexia | 1 year
Source localization of audio-visual integration processes | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Teija Kujala, Prof., Principal Investigator — Cognitive Brain Research Unit, Institute of Behavioural Sciences, University of Helsinki
Locations (1):
- Laboratory of CBRU, Institute of Behavioural Sciences, University of Helsinki, Helsinki, Uusimaa, Finland

REFERENCES:
- [Background] Dimitriadis SI, Laskaris NA, Simos PG, Micheloyannis S, Fletcher JM, Rezaie R, Papanicolaou AC. Altered temporal correlations in resting-state connectivity fluctuations in children with reading difficulties detected via MEG. Neuroimage. 2013 Dec;83:307-17. doi: 10.1016/j.neuroimage.2013.06.036. Epub 2013 Jun 15. PMID 23777755
- [Background] Giraud AL, Ramus F. Neurogenetics and auditory processing in developmental dyslexia. Curr Opin Neurobiol. 2013 Feb;23(1):37-42. doi: 10.1016/j.conb.2012.09.003. Epub 2012 Oct 3. PMID 23040541
- [Background] Hannula-Jouppi K, Kaminen-Ahola N, Taipale M, Eklund R, Nopola-Hemmi J, Kaariainen H, Kere J. The axon guidance receptor gene ROBO1 is a candidate gene for developmental dyslexia. PLoS Genet. 2005 Oct;1(4):e50. doi: 10.1371/journal.pgen.0010050. Epub 2005 Oct 28. PMID 16254601
- [Background] Hasson U, Nir Y, Levy I, Fuhrmann G, Malach R. Intersubject synchronization of cortical activity during natural vision. Science. 2004 Mar 12;303(5664):1634-40. doi: 10.1126/science.1089506. PMID 15016991
- [Background] Kere J. The molecular genetics and neurobiology of developmental dyslexia as model of a complex phenotype. Biochem Biophys Res Commun. 2014 Sep 19;452(2):236-43. doi: 10.1016/j.bbrc.2014.07.102. Epub 2014 Jul 28. PMID 25078623
- [Background] Kujala T, Karma K, Ceponiene R, Belitz S, Turkkila P, Tervaniemi M, Naatanen R. Plastic neural changes and reading improvement caused by audiovisual training in reading-impaired children. Proc Natl Acad Sci U S A. 2001 Aug 28;98(18):10509-14. doi: 10.1073/pnas.181589198. Epub 2001 Aug 21. PMID 11517333
- [Background] Kujala T, Lovio R, Lepisto T, Laasonen M, Naatanen R. Evaluation of multi-attribute auditory discrimination in dyslexia with the mismatch negativity. Clin Neurophysiol. 2006 Apr;117(4):885-93. doi: 10.1016/j.clinph.2006.01.002. Epub 2006 Feb 23. PMID 16497552
- [Background] Kujala T, Naatanen R. The mismatch negativity in evaluating central auditory dysfunction in dyslexia. Neurosci Biobehav Rev. 2001 Aug;25(6):535-43. doi: 10.1016/s0149-7634(01)00032-x. PMID 11595273
- [Background] Kujala T, Tervaniemi M, Schroger E. The mismatch negativity in cognitive and clinical neuroscience: theoretical and methodological considerations. Biol Psychol. 2007 Jan;74(1):1-19. doi: 10.1016/j.biopsycho.2006.06.001. Epub 2006 Jul 17. PMID 16844278
- [Background] Lankinen K, Saari J, Hari R, Koskinen M. Intersubject consistency of cortical MEG signals during movie viewing. Neuroimage. 2014 May 15;92:217-24. doi: 10.1016/j.neuroimage.2014.02.004. Epub 2014 Feb 12. PMID 24531052
- [Background] Leppanen PH, Richardson U, Pihko E, Eklund KM, Guttorm TK, Aro M, Lyytinen H. Brain responses to changes in speech sound durations differ between infants with and without familial risk for dyslexia. Dev Neuropsychol. 2002;22(1):407-22. doi: 10.1207/S15326942dn2201_4. PMID 12405511
- [Background] Lovio R, Halttunen A, Lyytinen H, Naatanen R, Kujala T. Reading skill and neural processing accuracy improvement after a 3-hour intervention in preschoolers with difficulties in reading-related skills. Brain Res. 2012 Apr 11;1448:42-55. doi: 10.1016/j.brainres.2012.01.071. Epub 2012 Feb 7. PMID 22364735
- [Background] Lovio R, Naatanen R, Kujala T. Abnormal pattern of cortical speech feature discrimination in 6-year-old children at risk for dyslexia. Brain Res. 2010 Jun 4;1335:53-62. doi: 10.1016/j.brainres.2010.03.097. Epub 2010 Apr 8. PMID 20381471
- [Background] Mittag M, Thesleff P, Laasonen M, Kujala T. The neurophysiological basis of the integration of written and heard syllables in dyslexic adults. Clin Neurophysiol. 2013 Feb;124(2):315-26. doi: 10.1016/j.clinph.2012.08.003. Epub 2012 Aug 30. PMID 22939780
- [Background] Naatanen R, Lehtokoski A, Lennes M, Cheour M, Huotilainen M, Iivonen A, Vainio M, Alku P, Ilmoniemi RJ, Luuk A, Allik J, Sinkkonen J, Alho K. Language-specific phoneme representations revealed by electric and magnetic brain responses. Nature. 1997 Jan 30;385(6615):432-4. doi: 10.1038/385432a0. PMID 9009189
- [Background] Naatanen R, Paavilainen P, Rinne T, Alho K. The mismatch negativity (MMN) in basic research of central auditory processing: a review. Clin Neurophysiol. 2007 Dec;118(12):2544-90. doi: 10.1016/j.clinph.2007.04.026. Epub 2007 Oct 10. PMID 17931964
- [Background] Naatanen R, Pakarinen S, Rinne T, Takegata R. The mismatch negativity (MMN): towards the optimal paradigm. Clin Neurophysiol. 2004 Jan;115(1):140-4. doi: 10.1016/j.clinph.2003.04.001. PMID 14706481
- [Background] Neuhoff N, Bruder J, Bartling J, Warnke A, Remschmidt H, Muller-Myhsok B, Schulte-Korne G. Evidence for the late MMN as a neurophysiological endophenotype for dyslexia. PLoS One. 2012;7(5):e34909. doi: 10.1371/journal.pone.0034909. Epub 2012 May 14. PMID 22606227
- [Background] Ramus F. Dyslexia. Talk of two theories. Nature. 2001 Jul 26;412(6845):393-5. doi: 10.1038/35086683. No abstract available. PMID 11473297
- [Background] Ramus F, Marshall CR, Rosen S, van der Lely HK. Phonological deficits in specific language impairment and developmental dyslexia: towards a multidimensional model. Brain. 2013 Feb;136(Pt 2):630-45. doi: 10.1093/brain/aws356. PMID 23413264
- [Background] Salmelin R. Clinical neurophysiology of language: the MEG approach. Clin Neurophysiol. 2007 Feb;118(2):237-54. doi: 10.1016/j.clinph.2006.07.316. Epub 2006 Sep 27. PMID 17008126
- [Background] Scerri TS, Schulte-Korne G. Genetics of developmental dyslexia. Eur Child Adolesc Psychiatry. 2010 Mar;19(3):179-97. doi: 10.1007/s00787-009-0081-0. Epub 2009 Nov 29. PMID 20091194
- [Background] Schulte-Korne G, Deimel W, Bartling J, Remschmidt H. Auditory processing and dyslexia: evidence for a specific speech processing deficit. Neuroreport. 1998 Jan 26;9(2):337-40. doi: 10.1097/00001756-199801260-00029. PMID 9507979
- [Background] Schumacher J, Anthoni H, Dahdouh F, Konig IR, Hillmer AM, Kluck N, Manthey M, Plume E, Warnke A, Remschmidt H, Hulsmann J, Cichon S, Lindgren CM, Propping P, Zucchelli M, Ziegler A, Peyrard-Janvid M, Schulte-Korne G, Nothen MM, Kere J. Strong genetic evidence of DCDC2 as a susceptibility gene for dyslexia. Am J Hum Genet. 2006 Jan;78(1):52-62. doi: 10.1086/498992. Epub 2005 Nov 17. PMID 16385449
- [Background] Shtyrov Y, Nikulin VV, Pulvermuller F. Rapid cortical plasticity underlying novel word learning. J Neurosci. 2010 Dec 15;30(50):16864-7. doi: 10.1523/JNEUROSCI.1376-10.2010. PMID 21159957
- [Background] Temple E. Brain mechanisms in normal and dyslexic readers. Curr Opin Neurobiol. 2002 Apr;12(2):178-83. doi: 10.1016/s0959-4388(02)00303-3. PMID 12015234
- [Background] Wolf M. Rapid alternating stimulus naming in the developmental dyslexias. Brain Lang. 1986 Mar;27(2):360-79. doi: 10.1016/0093-934x(86)90025-8. PMID 3513900
- [Background] Lyon, G.R. et al., 2003. Defining Dyslexia , Comorbidity , Teachers ' Knowledge of Language and Reading A Definition of Dyslexia. Annals of Dyslexia, 53(1), pp.1-14.
- [Background] Nevala, J., Kairaluoma, L. & Ahonen, T., 2006. Lukemis-ja kirjoittamistaitojen yksilötestistö nuorille ja aikuisille. Jyväskylä: Niilo Mäki
- [Background] Wechsler, D., 1997. Wechsler Adult Intelligence Scale (Third Edition), San Antonio, TX: The Psychological Corporation. Helsinki: Psykologien kustannus Oy.
- [Background] Wechsler, D., 1997. The Wechsler Memory Scale (Third Edition), San Antonio, TX: The Psychological Corporation. Helsinki: Psykologien kustannus Oy.
- See also: Suppanen, E., 2014. Inter-subject correlation of MEG data during movie viewing. Master's thesis, Aalto University School of Electrical Engineering. — http://urn.fi/URN:NBN:fi:aalto-201412303344
- See also: Thiede, A., 2014. Magnetoencephalographic (MEG) Inter-subject Correlation using Continuous Music Stimuli. Master's thesis, Aalto University School of Science. — http://urn.fi/URN:NBN:fi:aalto-201503061983